CLINICAL TRIAL: NCT04248374
Title: Fatty Acid Taste Rating With or Without Sour Taste Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Richard Mattes, Distinguished Professor, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 1907022413
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Taste, Altered
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Intervention Model Description: Fatty Acid taste with and without sour adaptation
Who Masked: Participant
Masking Description: three random number and covered sample cup[
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fatty Acid Taste (No Intervention): Fatty acid taste without sour adaptation
- Fatty Acid Taste after sour adaptation (Experimental): Fatty Acid Taste after sour adaptation
  Interventions: Other: Taste Intensity

INTERVENTIONS:
Other: Taste Intensity — Taste intensity with and without sour adaptation
  Arms: Fatty Acid Taste after sour adaptation

SUMMARY:
We are trying to figure out whether the fatty acid taste is differentiated from sour taste.

DETAILED DESCRIPTION:
Participants will be asked to provide general demographic information such as gender, age and ethnicity. Their height and weight will be measured. Then, they will be trained with one of the sample solutions for intensity rating and adaptation to sour taste. There will be eight different sample solutions containing sucrose esters, xanthan gums to help fatty acids stay dissolved, and either acetic acid for sour compounds or, butyric acid, caproic acid, caprylic acid, capric acid, lauric acid, oleic acid, or linoleic acid for fatty acid taste. 2 g of each palmitic acid and stearic acids in solid form (their melting points are above body temperature) will also be placed in participants' mouth. All of these compounds are common in the commercial food supply.

The study procedure entails two sets of taste intensity ratings without (Test A) or with (Test B) sour taste adaptation. For test A, participants will taste one of the eight solutions or one of solid fatty acids, and rate its intensity before and after expectorating it. They will not swallow any samples and they will rinse their tongues thoroughly with 1% ethanol solution and water after expectorating the solution. They will consume one piece of unsalted cracker and rinse their tongues thoroughly again. Before moving to the next step, they will be asked to describe the taste quality of the sample solution they just tasted. They will repeat this procedure with the rest of the sample solutions.

For test B, participants will follow the same procedure of taste intensity ratings but with sour taste adaptation. For sour taste adaptation, the participants will hold sour taste solutions in their mouth for 5 seconds and rate its taste intensity. They will repeat rating the sourness until they rate its intensity as less than weak. When they feel the sour taste solution weak, they will taste one of the eight solutions and repeat the intensity rating with one of the sample solutions. After the taste intensity rating, the participants will be asked to describe the taste quality of the sample solution they just tasted. They will repeat this procedure with the rest of the sample solutions.

The participants will do both test A and B twice in random order on two separate days. Taste testing is expected to take 1 hour each day. They will receive $20 at the end of the two test days as compensation for their participation.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* taste disorder no allergy to alcohol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Taste Intensity | 4 hours
  two sets of taste intensity ratings without (Test A) or with (Test B) sour taste adaptation. For test A, participants will taste one of the eight solutions or one of solid fatty acids, and rate its intensity before and after expectorating it.

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Mattes, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No